CLINICAL TRIAL: NCT06799429
Title: Implementing Brain Health Fitness: an On-going Individual Coaching and Exercise Intervention for People Living with Mild-moderate Cognitive Impairments in South Carolina
Brief Title: Brain Health Fitness Program: Exercise for People with Mild-moderate Cognitive Impairments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Foundation of Physical Therapy Research (Unknown)
Responsible Party: Principal Investigator, Elizabeth Regan, Associate Professor, University of South Carolina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00139826
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Cognitive Impairment
Keywords: cognitive impairment; exercise
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supervised In-Person Group (Experimental): For the in-person exercise group, exercise activity will be in the twice weekly in-person supervised, directed sessions at the Train Your Brain Fitness Center at the Arnold School of Public Health in Columbia, South Carolina. The exercise intervention will have a goal of up to120 minutes (60 minutes 2 x a week) of moderate intensity exercise, building up to that amount based on ability. This will include 45-60 minutes per week of cardiovascular activity (walking/jogging outside or on a treadmill, stationary bicycling (arm or traditional leg), rowing on an ergometer), 30-60 minutes of strength training (major muscle groups of the trunk, upper and lower extremities) and 15-30 minutes of balance, agility, and mobility exercises. Participants will ramp up to this level depending on their previous activity levels, and initial measures.
  Interventions: Behavioral: Supervised in-person group
- Monitored Distance Group (Experimental): For the monitored distance group, all activities will be performed at home or in a public gym environment near their home with prescribed plan provided by a fitness coach. The exercise intervention will have a goal of up to 120 minutes (60 minutes 2 x a week) of moderate intensity exercise, building up to that amount based on ability. This will include 45-60 minutes per week of cardiovascular activity (walking/jogging outside or on a treadmill, stationary bicycling (arm or traditional leg), rowing on an ergometer), 30-60 minutes of strength training (major muscle groups of the trunk, upper and lower extremities) and 15-30 minutes of balance, agility, and mobility exercises. Participants will ramp up to this level depending on their previous activity levels, and initial measures.
  Interventions: Behavioral: Monitored distance group

INTERVENTIONS:
Behavioral: Supervised in-person group — Individually prescribed and directed/supervised by a fitness trainer in-person, multi-mode exercise 2 x a week for 30-60 minutes The fitness trainer is with the participant while they exercise.
  Arms: Supervised In-Person Group
Behavioral: Monitored distance group — Individually prescribed ulti-mode exercise 2 x a week for 30-60 minutes. Written plan/feedback and support by phone/text or email is provided by a fitness trainer who is not present with the participant when they exercise.
  Arms: Monitored Distance Group

SUMMARY:
The goal of this clinical trial is to test a 6-month, twice a week, moderate intensity exercise and coaching program (an in-person group and a distance group) for adults with mild-moderate cognitive impairments living in South Carolina. The main questions it aims to answer are:

1. Is the program practical to conduct, and it is acceptable and enjoyable? The hypothesis is that it will be possible to recruit participants, obtain the desired dosage of moderate intensity fitness and strength training twice a week.
2. Are their changes at 3-months and 6-months in endurance, mobility, cognitive function and perception of cognitive function? The hypotheses are that endurance, strength and mobility will improve and cognitive measures will not decline (remain the same or improve).

Participants will exercise twice a week in-person with a coach or at a distance location with coaching support for six months.

DETAILED DESCRIPTION:
In person Exercise Group:

The exercise program interventions will be individualized based on exercise history, and initial assessments by the primary investigator (a physical therapist). The program will focus on building up to 30 minutes of moderate intensity endurance activity and up to 30 minutes of strength training, balance training and mobility training. Participants will attend times per week for six months. Coaches will provide exercise plans, and monitor and provide feedback as participants exercise. Participants will wear a heart rate monitor to record exertion. Participants will be able to continuously attend as long as they are attending regularly.

Distance Exercise Group:

The exercise program interventions will be individualized based on exercise history, and initial assessments by the primary investigator (a physical therapist) which will occur in person. The program will focus on building up to 30 minutes of moderate intensity endurance activity and up to 30 minutes of strength training, balance training and mobility training. Participants will exercise on their own 2 x a week for 6 months.Coaches will prescribe an exercise program that can be performed at a local fitness facility or at home and it will be shared through a coaching software. Participants will log their exercises either in the coaching software or in paper formats, have weekly check-ins with fitness center coaches and have options to message the fitness center coaches with questions. Participants who do not log any activity and miss weekly check-ins will have follow up from fitness center coaches.

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of mild-moderate cognitive impairment
* medically cleared for exercise
* able to follow 2-step commands Exclusion criteria are significant pain with movement (>5/10)

Exclusion Criteria:

* significant pain with movement (>5/10)
* severe balance impairments or lack of independence on and off exercise equipment (by physical therapist judgement).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Aim 1 Feasibility: Recruitment and Uptake through qualified referrals | through study completion, an average of 1 year
  percent of qualified referrals beginning the program
Aim 1 Feasibility: Program Fidelity Dosage: session adherence | through study completion, an average of 1 year
  mean percentage adherence (number of sessions completed / number of sessions scheduled)
Aim 1 Feasibility: Program Fidelity Dosage: Session Duration | through study completion, an average of 1 year
  mean percentage duration
Aim 1 Feasibility: Program Fidelity: Exercise Intensity | through study completion, an average of 1 year
  mean percent of time spent in target heart rate zone of 60-85% of age predicted maximum
Aim 1 Feasibility: Acceptability: Participant Satisfaction | through study completion, an average of 1 year
  mean of 5 point likert scale 1-not satisfied to 5-extremely satisfied
Aim 2 Exploratory Individual Outcomes: Processing Speed and Executive Function through the Oral Symbol Digits Test (NIH Toolbox) | pre-program (baseline), mid-program (3 months) and post-program (6-months)
  Score is number of correct responses (0-144), with higher score as better performance
Aim 2 Exploratory Individual Outcomes: Cardiovascular Endurance through the six-minute walk test | pre-program (baseline), mid-program (3 months) and post-program (6-months)
  Score is meters walked, higher is better performance

SECONDARY OUTCOMES:
Aim 2 Exploratory Individual Outcomes: Mobility and Balance through the Short Physical Performance Battery | pre-program (baseline), mid-program (3 months) and post-program (6-months)
  Score is 0-12 with higher as better performance
Aim 2 Exploratory Individual Outcomes: Grip Strength using a hand-held grip dynamometer (lbs. of force) | pre-program (baseline), mid-program (3 months) and post-program (6-months)
  Measured bilateral in lbs of force, higher is better performance
Aim 2 Exploratory Individual Outcomes: Perception of cognition through the Patient-Reported Outcomes Measurement Information System (PROMIS) Computer Adaptive Testing survey | pre-program (baseline), mid-program (3 months) and post-program (6-months)
  0-100% with lower than 50% below average and higher above average performance

CONTACTS AND LOCATIONS:
Locations (1):
- Arnold School of Public Health, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic, clinical data, outcomes data (survey and functional measures) and exercise intervention session data (mode, intensity, duration) will be generated for all participants. Demographic and clinical data will be collected at the start of the intervention. Outcomes data will be collected at the beginning of the program, at mid-point (3 months) and at the end of the program (6 months). All data will be de-identified prior to receipt by the data archive repository, but information to tie each participant to a unique identifier for the data archive will be maintained for each participant.
  In addition, global program feasibility data (recruitment and uptake, fidelity, intensity, acceptability) will be generated.